CLINICAL TRIAL: NCT02506660
Title: Interscalene Block With Low-dose IV vs. Perineural Dexamethasone for Shoulder Arthroscopy
Acronym: Dex ISB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-379
Record Dates: First submitted 2015-07-02; First posted 2015-07-23 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Pain; Shoulder Arthroscopy
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Intravenous dexamethasone (Active Comparator): Patients will receive 1 cc (1 mg) dexamethasone intravenously and a block containing 15 cc bupivacaine 0.5% and 1 cc saline.
  Interventions: Drug: Bupivacaine; Drug: Intravenous dexamethasone; Drug: Perineural saline
- Perineural dexamethasone (Experimental): Patients will receive 1 cc saline intravenously and a block containing 15 cc bupivacaine 0.5% and 1 cc (1 mg) dexamethasone.
  Interventions: Drug: Bupivacaine; Drug: Perineural dexamethasone; Drug: Intravenous saline

INTERVENTIONS:
Drug: Bupivacaine
Drug: Perineural dexamethasone — Dexamethasone in nerve block
  Arms: Perineural dexamethasone
Drug: Intravenous dexamethasone
  Arms: Intravenous dexamethasone
Drug: Intravenous saline
  Arms: Perineural dexamethasone
Drug: Perineural saline — Saline in nerve block
  Arms: Intravenous dexamethasone

SUMMARY:
Many patients undergoing ambulatory shoulder arthroscopy experience moderate to severe pain after surgery. Finding ways to minimize postoperative pain are ideal. Dexamethasone is a corticosteroid that is commonly used to prevent and/or treat nausea and inflammation. The addition of higher doses of dexamethasone to nerve blocks, which are injections of local anesthetics into the upper shoulder area, has been shown to prolong block duration and reduce pain. However, it is unclear whether the advantage of longer pain relief outweighs patient dissatisfaction with the prolonged feeling of a numb arm. Furthermore, recent studies have shown that systemic, intravenously administered dexamethasone may similarly reduce pain levels when compared with dexamethasone in the block. In our study, the investigators propose to examine the effect of low-dose IV versus block dexamethasone on interscalene block duration in patients undergoing shoulder arthroscopy. Most studies have used 4 mg or more. One study suggests that 1 mg may have the same effect as larger doses. Our aims are to determine whether the addition of low-dose dexamethasone to a local anesthetic in the block can prolong its duration, and whether there are differences in postoperative pain, consumption of painkillers, side effects, and satisfaction in patients who received IV or block dexamethasone. Patients (128 total) will be randomly assigned to either receive IV or block dexamethasone, and postoperative assessments (pain, painkiller use, side effects, block duration, satisfaction, complications) will be made via phone at 2, 3, 4 (if needed), and 7-10 days after surgery. Results from this study will reveal whether patients prefer the longer-duration analgesia that may be obtained with low-dose dexamethasone in the block.

ELIGIBILITY:
Inclusion Criteria:

* Patients having ambulatory arthroscopic shoulder surgery under ultrasound-guided interscalene block (rotator cuffs, acromioplasties, stabilizations, labral repairs, etc.)
* Age 18-70 years

Exclusion Criteria:

* Contraindication to interscalene block
* Known allergy/sensitivity to any study medications
* Having taken daily steroids for 10 days or longer anytime during the past year
* Body mass index <18 or >40
* History of uncontrolled nausea and vomiting with opioids or severe post-op nausea and vomiting (to prevent any need for higher doses of IV dexamethasone)
* Non-English speaking
* Revision procedures
* Additional procedures (e.g., removal of hardware, procedures involving other areas, etc.)
* Planned open procedures
* History of diabetes
* Arthroscopic irrigation and debridement secondary to infection
* Peripheral neuropathies affecting the operative extremity
* Having taken opiates daily for 10 days or longer immediately preceding surgery, 3 times a week for greater than 3 months anytime in the past year, or currently taking for anything other than shoulder pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kahn, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] Kahn RL, Cheng J, Gadulov Y, Fields KG, YaDeau JT, Gulotta LV. Perineural Low-Dose Dexamethasone Prolongs Interscalene Block Analgesia With Bupivacaine Compared With Systemic Dexamethasone: A Randomized Trial. Reg Anesth Pain Med. 2018 Aug;43(6):572-579. doi: 10.1097/AAP.0000000000000817. PMID 29889698

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Dexamethasone: Patients will receive 1 cc (1 mg) dexamethasone intravenously and a block containing 15 cc bupivacaine 0.5% and 1 cc saline.
  Bupivacaine
  Intravenous dexamethasone
  Perineural saline: Saline in nerve block
- Perineural Dexamethasone: Patients will receive 1 cc saline intravenously and a block containing 15 cc bupivacaine 0.5% and 1 cc (1 mg) dexamethasone.
  Bupivacaine
  Perineural dexamethasone: Dexamethasone in nerve block
  Intravenous saline
Period: Overall Study
Arm/Group | Intravenous Dexamethasone | Perineural Dexamethasone
Started | 64 | 64
Completed | 62 | 63
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Dexamethasone | Perineural Dexamethasone | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (14.6) | 49.9 (13.6) | 48.3 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 39 | 37 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 57 | 57 | 114
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Nerve Block Duration
Description: Time at which the pain relief from the block has completely worn off
Time Frame: Postoperative day 2+
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Intravenous Dexamethasone | Perineural Dexamethasone
Number analyzed (Participants) | 62 | 63
Hours | 22.2 [19.5 to 26] | 25.7 [22.2 to 31.5]

2. Secondary Outcome: Numerical Rating Scale Pain Scores
Description: The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Time Frame: Duration of stay in recovery room after surgery (average of 3 hours)
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Intravenous Dexamethasone | Perineural Dexamethasone
Number analyzed (Participants) | 62 | 63
Units on a Scale | 0 [0 to 2] | 0 [0 to 2]

3. Secondary Outcome: Opioid Consumption
Time Frame: Postoperative day 2, postoperative day 3
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intravenous Dexamethasone | Perineural Dexamethasone
Number analyzed (Participants) | 62 | 63
mg
  Postoperative day 2 | 67.3 (55.7) | 67.4 (51)
  postoperative day 3 | 33 (48.6) | 39.7 (55.3)

4. Secondary Outcome: Side Effects
Description: Opioid-related symptom distress scale is calculated using responses to the symptom severity questions only.
  For each symptom, severity is assessed by the question: "(If yes), how severe was it usually?" (In the past 24 hours) The responses to the severity questions are measured on a 5-point scale from 0-4 in ascending order as follows: Did not have symptom (0) Slight (1) Moderate (2) Severe (3) Very severe (4)
Time Frame: Postoperative day 2, postoperative day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Dexamethasone | Perineural Dexamethasone
Number analyzed (Participants) | 60 | 63
units on a scale
  Postoperative day 2 | 0.5 (0.5) | 0.6 (0.5)
  postoperative day 3 | 0.4 (0.4) | 0.4 (0.4)

5. Secondary Outcome: Block Satisfaction
Description: 0-10 scale (0=not satisfied; 10=extremely satisfied)
Time Frame: Postoperative day 2, postoperative day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Dexamethasone | Perineural Dexamethasone
Number analyzed (Participants) | 58 | 61
units on a scale
  postoperative day 2 | 8.1 (2.2) | 8.1 (2.2)
  postoperative day 3 | 8.0 (2.1) | 7.5 (2.5)

6. Secondary Outcome: Block-related Complications
Time Frame: Postoperative day 7-10
Measure: Number; unit: patients with block complications
Arm/Group | Intravenous Dexamethasone | Perineural Dexamethasone
Number analyzed (Participants) | 62 | 63
patients with block complications | 0 | 0

7. Secondary Outcome: % of Participants Who Guessed the Correct Group
Description: Patients will be asked whether they believe they were in the IV dexamethasone or intravenous dexamethasone group
Time Frame: Postoperative day 7-10
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Intravenous Dexamethasone | Perineural Dexamethasone
Number analyzed (Participants) | 57 | 56
% of participants | -7 [-16 to 2] | 3.4 [-6.3 to 13.2]

ADVERSE EVENTS:
Arm/Group | Intravenous Dexamethasone | Perineural Dexamethasone
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 0/62 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes